CLINICAL TRIAL: NCT04406961
Title: A Randomized Controlled Trial Comparing Antegrade Sphincterotomy Dovbenko (ASD) With Conventional Pull-Type Sphincterotomy in Patients Undergoing ERCP
Brief Title: Endoscopic Antegrade Sphincterotomy (ASD) Versus Standard Sphincterotomy
Acronym: ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Medical Clinical Center of the Southern Region, Ukraine (Other)
Responsible Party: Principal Investigator, Oleg Dovbenko, MD, Head of the Department of Endoscopic Surgery, Military Medical Clinical Center of the Southern Region, Military Medical Clinical Center of the Southern Region, Ukraine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol-273; 273 (Other: Bioethics Committee of the National Academy of Sciences of Ukraine)
Record Dates: First submitted 2020-05-02; First posted 2020-05-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Choledocholithiasis; Papillary Stenosis; Biliary Obstruction; Gallstone Disease; External Biliary Fistula; Malignant Biliary Obstruction; Benign Biliary Strictures With Current or Prior Biliary Obstruction
Keywords: endoscopic transpapillary antegrade sphincterotomy (ASD); antegrade sphincterotome; preservation of the function of the sph. of Oddi; avoid cholecystectomy
MeSH Terms: conditions — Choledocholithiasis; Cholelithiasis | interventions — Sphincterotomy, Endoscopic

STUDY DESIGN:
Intervention Model Description: This parallel-group, randomized controlled trial compares two endoscopic sphincterotomy techniques in patients undergoing transpapillary interventions: (1) conventional pull-type endoscopic sphincterotomy (EST), and (2) antegrade sphincterotomy developed by Dr. Dovbenko (Antegrade Sphincterotomy Dovbenko, ASD), which selectively incises only the circular muscle layer of the sphincter of Oddi using a dedicated sphincterotome (Ukrainian Patent No. UA 117987C2, 2019). The primary analysis evaluates the relative risk and 95% confidence interval for procedure-related complications, including bleeding, perforation, post-ERCP pancreatitis, and need for cholecystectomy.
Masking Description: Due to the nature of the endoscopic surgical interventions, neither participants nor investigators (including endoscopists and treating physicians) could be blinded to treatment allocation. All outcomes were assessed using standardized, objective criteria as defined in the European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline on post-ERCP complications (2023) and the ESGE Technical Guideline on endoscopic sphincterotomy (2020).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard sphincterotomy. (Active Comparator): Patients in this group underwent conventional retrograde endoscopic sphincterotomy using a standard Erlangen-type "pull" sphincterotome. Following deep biliary cannulation, the sphincterotome was used to perform a standard pull-type incision across the major duodenal papilla. In 20% of cases, a needle-knife precut papillotomy was performed to facilitate biliary access. A total of 760 patients were enrolled in this arm. Procedure-related complications were prospectively recorded, including: post-ERCP pancreatitis, bleeding, perforation, cholangitis, acute cholecystitis, recurrent choledocholithiasis, and papillary restenosis.
  Interventions: Procedure: Endoscopic sphincterotomy.; Device: The standard sphincterotome.
- Antegrade Sphincterotomy Dovbenko (ASD) (Experimental): Patients underwent endoscopic transpapillary antegrade sphincterotomy (Antegrade Sphincterotomy Dovbenko, ASD) using a dedicated sphincterotome designed by Dr. Dovbenko (Ukrainian Patent No. UA 117987C2, 2019). Following deep biliary cannulation, the sphincterotome was advanced transpapillary and used to perform an antegrade incision selectively targeting only the circular muscle layer of the sphincter of Oddi, with preservation of the longitudinal layer and duodenal integrity. In 20% of cases, needle-knife precut papillotomy was performed to facilitate initial biliary cannulation.
  Interventions: Procedure: Endoscopic transpapillary antegrade sphincterotomy developed by Dr. Dovbenko.; Device: The antegrade sphincterotome developed by Dr. Dovbenko.

INTERVENTIONS:
Procedure: Endoscopic transpapillary antegrade sphincterotomy developed by Dr. Dovbenko. — Sph. Oddi consists of a longitudinal and circular smooth muscle layers. Circular muscle fibers form the pancreatic and duodenal parts. Anatomical justification was cutting of only the circular layer of sph Oddi by special sphincterotome. Papillary stenosis and stenosis terminal part of common bile duct due to damage only circular layer sph Oddi. Anterograde direction and hooked form of sphincterotome (endoscopic antegrade sphincterotomy- ASD) allows to capture only need layer and control depth. Also ASD was performed patient with SOD (I-III) with preservation of the longitudinal muscular layer sph Oddi and septum of papilla.
  Other Names: ASD
  Arms: Antegrade Sphincterotomy Dovbenko (ASD)
Device: The antegrade sphincterotome developed by Dr. Dovbenko. — A device is represented by a teflon catheter in the distal part of which a double tube of variable shape is created. The proximal part of the ASD sphincterotome consists of a handle, and a metal wire is located inside the teflon catheter for connection to an electrosurgical unit. On the distal part, the teflon catheter is formed of a double tube length is 10 to 35 mm. The metal wire exits the catheter at a distance 10 to 35 mm from the tip and enters into the tip the second teflon tube. The distal part of the knife is formed shape a hook. A metal cutting wire is located between two tubes. Moving the handle the metal wire is shifted. Pushing the metal wire or approaching in the distal part the second tube sets the depth of cut. The incision is made by moving on guidewire in bile duct. The power settings vary.
  Arms: Antegrade Sphincterotomy Dovbenko (ASD)
Procedure: Endoscopic sphincterotomy. — Endoscopic standard sphincterotomy aims at opening bile duct or pancreatic duct by cutting the papilla and sphincter muscles. After deep bile duct cannulation, the standard sphincterotome is retracted until one fourth to one half of the wire length is exposed outside the papilla. The sphincterotome is slightly bowed so that the wire is in contact with the roof. The incision is made lifting the sphincterotome against the papillary roof using the elevator and up-down controls while applying short bursts of current. The power settings vary. The extent of the sphincterotomy is limited by the length of the intraduodenal portion of the common bile duct.
  Arms: Standard sphincterotomy.
Device: The standard sphincterotome. — The standard sphincterotome, the Erlangen "pull-type" model, consists of a catheter containing a cautery wire exposed 15 to 25 mm near the tip of the instrument. The leading tip distal to the wire, the "nose," is 5 to 10 mm in diameter. After deep bile duct cannulation, the sphincterotome is retracted slowly, until one fourth to one half of the wire length is exposed outside the papilla. The sphincterotome is slightly bowed so that the wire is in contact with the roof. The incision is made by lifting the sphincterotome against the papillary roof using the elevator and up-down controls while applying short bursts of current. The power settings vary.
  Other Names: "pull-type" model, the Erlangen.
  Arms: Standard sphincterotomy.

SUMMARY:
This study compares endoscopic transpapillary antegrade sphincterotomy developed by Dr. Dovbenko (Antegrade Sphincterotomy Dovbenko, ASD) with conventional pull-type endoscopic sphincterotomy (EST) in patients undergoing transpapillary interventions for various indications, including biliary stone disease, major duodenal papilla stenosis, choledocholithiasis, and other conditions requiring access to the biliary and/or pancreatic ducts. The ASD technique is performed using a dedicated sphincterotome designed by Dr. Dovbenko. Both the technique and the device are patented in Ukraine (Patent No. UA 117987C2, 2019). This instrument enables selective incision of only the circular muscle layer of the sphincter of Oddi, thereby preserving its sphincteric function and minimizing trauma to the duodenal wall. The primary objective of the study is to evaluate the relative risk of procedure-related complications, including bleeding, perforation, post-ERCP pancreatitis, and the need for cholecystectomy.

DETAILED DESCRIPTION:
Anatomical studies confirm that the sphincter of Oddi comprises an inner circular muscle layer, functionally and structurally distinct from the duodenum, and an outer longitudinal layer derived from the duodenal wall. Preservation of this architecture is critical to maintaining sphincteric function. Standard pull-type sphincterotomy frequently disrupts both layers and adjacent duodenal tissue, contributing to procedure-related complications in up to 23% of ERCPs, including bleeding (≤3%), perforation (≤1%), and post-sphincterotomy reflux complications.

Antegrade Sphincterotomy Dovbenko (ASD) was developed to address these limitations. Using a dedicated sphincterotome (Ukrainian Patent No. UA 117987C2, 2019), ASD enables selective incision of the circular layer while sparing the longitudinal layer and duodenal integrity.

This prospective, randomized, parallel-group trial (NCT04406961) enrolled 1,521 patients requiring transpapillary intervention for biliary or pancreatic indications. Patients were assigned to ASD (n=761) or conventional EST (n=760).

In the ASD group, a trend toward reduced major complications was observed (RR 0.55; 95% CI 0.18-1.67); however, this difference did not reach statistical significance, likely due to the low absolute number of events. Notably, cholecystectomy was avoided in 71.2% of ASD patients with gallstone disease, compared to approximately 10% in the EST group. Temporary stenting (5-10 days) was used selectively to manage post-procedural edema. ASD should be performed exclusively by endoscopists with advanced transpapillary expertise.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Gallstone Disease. Must have anatomy of the esophagus of the stomach and duodenum for the introduction of a duodenoscope to the major duodenal papilla.

Exclusion Criteria:

The acute form of viral hepatitis of any etiology. Acute decompensated heart failure complicated by respiratory failure.

Ages: 18 Years to 102 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1521 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2025-12-21 (Actual)

PRIMARY OUTCOMES:
Composite incidence of major procedure-related adverse events | Up to 30 days after the procedure.
  Proportion of participants experiencing at least one of the following within 30 days: (1) post-ERCP pancreatitis (serum lipase ≥3× upper limit of normal plus abdominal pain persisting ≥24 hours requiring prolonged or unplanned hospitalization); (2) clinically significant bleeding (hemoglobin drop ≥2 g/dL and/or need for endoscopic, radiological, or surgical intervention); (3) duodenal or biliary perforation confirmed by imaging or surgery.

SECONDARY OUTCOMES:
Incidence of papillary restenosis requiring re-intervention | From 6 months to 5 years after the procedure
  Papillary restenosis is defined as recurrent biliary obstruction confirmed by imaging (CT, MRI, or cholangiography), characterized by:
  1. common bile duct diameter >11 mm, and
  2. total bilirubin >60 µmol/L (≈3.5 mg/dL) in the absence of other causes of obstruction.
  Only cases requiring endoscopic, radiological, or surgical re-intervention are counted as events.
Incidence of post-ERCP pancreatitis. | Within 72 hours after the procedure
  Post-ERCP pancreatitis is defined as new-onset abdominal pain persisting for at least 24 hours plus serum lipase level at least 3 times the upper limit of normal, requiring prolonged or unplanned hospitalization for pain management and monitoring.
Incidence of duodenal or biliary perforation. | From the start of the procedure up to 30 days after.
  Perforation is defined as a full-thickness defect of the duodenal or bile duct wall, confirmed by: (1) extraluminal contrast on cholangiography or fluoroscopy, (2) free air on abdominal X-ray or CT scan, or (3) intraoperative diagnosis. Perforations are classified as periampullary, duodenal, or biliary.
Incidence of clinically significant post-sphincterotomy bleeding | From the start of the procedure up to 30 days after
  Clinically significant bleeding is defined as: (1) a decrease in hemoglobin level of ≥2 g/dL from pre-procedure baseline, and/or (2) requirement for endoscopic, radiological, or surgical intervention to achieve hemostasis. Minor oozing not requiring intervention is not counted as an event.
Rate of cholecystectomy within 12 months | From the date of the procedure up to 12 months
  Proportion of participants with concomitant gallstone disease who undergo cholecystectomy within 12 months following the index ERCP procedure, regardless of symptoms. Only elective or urgent cholecystectomies performed for biliary pathology are included; procedures for unrelated indications are excluded.
Technical success: complete bile duct stone clearance | During the procedure
  Defined as the absence of residual filling defects in the common bile duct on post-procedure cholangiography (intraoperative or fluoroscopic). Clearance is confirmed before the end of the index ERCP session.
Need for repeat ERCP within 30 days | From the date of the index procedure up to 30 days after
  Proportion of participants requiring a repeat endoscopic retrograde cholangiopancreatography (ERCP) within 30 days after the index procedure due to: (1) incomplete stone clearance, (2) recurrent biliary obstruction, (3) post-procedure complications (e.g., cholangitis, bleeding, or stent dysfunction), or (4) other biliary or pancreatic indications directly related to the initial intervention.
  Elective ERCP for unrelated reasons is excluded.

CONTACTS AND LOCATIONS:
Locations (1):
- Oleg Dovbenko, Odesa, Odesa Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) collected during the trial, including de-identified baseline characteristics, procedural details, outcomes, and adverse events, will be available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD and supporting documents will be available beginning 3 months after publication of the primary results manuscript and will remain accessible for 5 years.
Access Criteria: Researchers may request access to de-identified IPD for non-commercial, scientifically valid research purposes. Requests must be submitted in writing to the Principal Investigator and will be reviewed by the Data Access Committee. Approved researchers will sign a data use agreement ensuring confidentiality and prohibiting re-identification.

REFERENCES:
- [Derived] Dovbenko O, Herasymenko O. Endoscopic management of hepaticojejunal anastomosis fistula after Whipple's resection. Endoscopy. 2024 Dec;56(S 01):E72-E73. doi: 10.1055/a-2226-0276. Epub 2024 Jan 23. No abstract available. PMID 38262462
- See also: Endoscopic transpapillary antegrade sphincterotomy (ASD): preliminary results. Endoscopy 2019;51(S 04):S192. Abstract presented at ESGE Days 2019, Prague. — https://doi.org/10.1055/s-0039-1681738
- See also: Diathermic knife and method of endoscopic transpapillary antegrade sphincterotomy developed by Dr. O.V. Dovbenko. Ukrainian Patent UA117987C2, issued 2018 — https://patents.google.com/patent/UA117987C2